CLINICAL TRIAL: NCT02018562
Title: Prospective Evaluation of a Tracheostomy Tube That Enables Communication in Ventilator Dependent Patients - A Pilot Study
Brief Title: Evaluation of a Tracheostomy Tube That Enables Communication
Acronym: BLUSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00086689
Record Dates: First submitted 2013-12-03; First posted 2013-12-23 (Estimated); Results first posted 2018-04-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Evaluate the Effect of a Talking Tracheostomy Tube on Quality of Life
Keywords: Quality of Life; Talking Tracheostomy Tube; Speech; Mechanically ventilated patients
MeSH Terms: conditions — Speech

STUDY DESIGN:
Masking Description: Unable to mask because patients and care providers were able to visualize the type of tracheostomy tub that was used.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): 1. The talking tracheostomy trial involves placement of a talking tracheostomy tube (Portex Blueline Ultra Suctionaid Tracheostomy Tube) by respiratory therapist after obtaining an order from an authorized prescriber (Physician or Nurse Practitioner). The Speech-Language Pathologist (SLP) sets up the tracheostomy tube for speech and then determines the optimal air flow required for voicing. This amount of air flow is communicated to the ICU staff for further use.
  2. We will ensure that the SLP meets with the patient for a minimum of 3 sessions within a week to optimize the use of a talking tracheostomy tube.
  i. SLP will also assess the duration of successful speech during each session
  ii. Sentence intelligibility will also be assessed during the 3rd session. This session will be audio-taped and reviewed by a second rater for sentence intelligibility.
  iii. SLP will determine the level of independence with talking tracheostomy during the 3rd session.
  Interventions: Device: Portex Blueline Ultra Suctionaid Tracheostomy Tube
- Control (No Intervention): This group will also receive talking tracheostomy tube trial as standard of care but a week later after the pre and post assessments have been completed

INTERVENTIONS:
Device: Portex Blueline Ultra Suctionaid Tracheostomy Tube
  Arms: Intervention

SUMMARY:
Verbal communication is vital to critically ill mechanically ventilated patient's quality of life (Hess, 2005). Patients who have a tracheostomy tube may be able to communicate using a speaking valve, however, some patients may not be able to tolerate cuff deflation for use of speaking valve. There are talking tracheostomy tubes that do not require cuff deflation to facilitate speech in this population. Unfortunately, not all candidates are offered these options due to lack of awareness. Recently, at our institution, there has been an increase in the use of these tubes to facilitate speech. One of the talking tracheotomy tubes that has proven to be effective is the Portex Blueline Ultra Suctionaid (BLUSA).

In 2010, we conducted a retrospective review of 4 cases and found that BLUSA tracheostomy helped facilitate communication in this unique population (IRB #: NA_00041547). We would now like to formally conduct a prospective pilot study to evaluate the feasibility of measuring outcomes of patients with a BLUSA using a pretest-posttest research design.

Communication empowers patients and allows healthcare staff to obtain a more accurate assessment of patients' condition and tailor care accordingly. Identifying the predictors of speech intelligibility and the impact of BLUSA on quality of life will promote communication between patients and healthcare providers.

Study Hypothesis: Determine the impact of a talking tracheostomy tube on quality of life in patients requiring prolonged mechanical ventilation in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated via tracheostomy
* Awake, alert, and attempting to communicate
* Able to understand English

Exclusion Criteria:

* Delirium
* Fresh tracheostomy within 48 hours
* Laryngectomy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-02-21 (Actual); Study Completion 2017-05-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Batty S. Communication, swallowing and feeding in the intensive care unit patient. Nurs Crit Care. 2009 Jul-Aug;14(4):175-9. doi: 10.1111/j.1478-5153.2009.00332.x. PMID 19531034
- [Background] Frost SA, Azeem A, Alexandrou E, Tam V, Murphy JK, Hunt L, O'Regan W, Hillman KM. Subglottic secretion drainage for preventing ventilator associated pneumonia: a meta-analysis. Aust Crit Care. 2013 Nov;26(4):180-8. doi: 10.1016/j.aucc.2013.03.003. Epub 2013 Apr 11. PMID 23583261
- [Background] Hess DR. Facilitating speech in the patient with a tracheostomy. Respir Care. 2005 Apr;50(4):519-25. PMID 15807915
- [Background] Husain T, Gatward JJ, Harris RD. Use of subglottic suction port to enable verbal communication in ventilator-dependent patients. Am J Respir Crit Care Med. 2011 Aug 1;184(3):384. doi: 10.1164/ajrccm.184.3.384. No abstract available. PMID 21804129
- [Result] Coffman HM, Rees CJ, Sievers AE, Belafsky PC. Proximal suction tracheotomy tube reduces aspiration volume. Otolaryngol Head Neck Surg. 2008 Apr;138(4):441-5. doi: 10.1016/j.otohns.2007.11.013. PMID 18359351
- [Result] Hofhuis JG, Spronk PE, van Stel HF, Schrijvers AJ, Rommes JH, Bakker J. Experiences of critically ill patients in the ICU. Intensive Crit Care Nurs. 2008 Oct;24(5):300-13. doi: 10.1016/j.iccn.2008.03.004. Epub 2008 May 9. PMID 18472265
- [Result] Lacherade JC, De Jonghe B, Guezennec P, Debbat K, Hayon J, Monsel A, Fangio P, Appere de Vecchi C, Ramaut C, Outin H, Bastuji-Garin S. Intermittent subglottic secretion drainage and ventilator-associated pneumonia: a multicenter trial. Am J Respir Crit Care Med. 2010 Oct 1;182(7):910-7. doi: 10.1164/rccm.200906-0838OC. Epub 2010 Jun 3. PMID 20522796
- [Result] Nomori H. Tracheostomy tube enabling speech during mechanical ventilation. Chest. 2004 Mar;125(3):1046-51. doi: 10.1378/chest.125.3.1046. PMID 15006967
- [Result] Pandian V, Maragos C, Turner L, Mirski M, Bhatti N, Joyner K. Model for best practice: nurse practitioner facilitated percutaneous tracheostomy service. ORL Head Neck Nurs. 2011 Spring;29(2):8-15. PMID 21675700
- [Result] Pandian V, Miller CR, Mirski MA, Schiavi AJ, Morad AH, Vaswani RS, Kalmar CL, Feller-Kopman DJ, Haut ER, Yarmus LB, Bhatti NI. Multidisciplinary team approach in the management of tracheostomy patients. Otolaryngol Head Neck Surg. 2012 Oct;147(4):684-91. doi: 10.1177/0194599812449995. Epub 2012 Jun 5. PMID 22675004
- [Derived] Pandian V, Cole T, Kilonsky D, Holden K, Feller-Kopman DJ, Brower R, Mirski M. Voice-Related Quality of Life Increases With a Talking Tracheostomy Tube: A Randomized Controlled Trial. Laryngoscope. 2020 May;130(5):1249-1255. doi: 10.1002/lary.28211. Epub 2019 Aug 6. PMID 31385620

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: 1. This involves placement of a talking tracheostomy tube (Portex Blueline Ultra Suctionaid Tracheostomy Tube) by respiratory therapist after obtaining an order from an authorized prescriber (Physician or Nurse Practitioner). The Speech-Language Pathologist (SLP) sets up the tracheostomy tube for speech and then determines the optimal air flow required for voicing. This amount of air flow is communicated to the ICU staff for further use.
  2. We will ensure that the SLP meets with the patient for a minimum of 3 sessions within a week to optimize the use of a talking tracheostomy tube.
  i. SLP will also assess the duration of successful speech during each session. ii. Sentence intelligibility will also be assessed during the 3rd session. This session will be audio-taped and reviewed by a second rater for sentence intelligibility.
  iii. SLP will determine the level of independence with talking tracheostomy during the 3rd session.
  Portex Blueline Ultra Suctionaid Tracheostomy Tube
Period: Overall Study
Arm/Group | Intervention | Control
Started | 25 | 25
Completed | 22 | 25
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Discharged prior to study completion | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.72 (17.47) | 57.92 (14.91) | 54.32 (16.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 10 | 15 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 25 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 9 | 18
  White | 14 | 16 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life
Description: Quality of Life in Mechanically Ventilated Patients Questionnaire (QOL-MV) was used to measure quality of life. It is a 12-item scale with each items 0 - 10 and total score ranges from 0 - 120. Lower scores refers to lower quality of life and Higher scores refer to higher level quality of life. To be assessed at baseline and 2 weeks post Portex Blueline Ultra Suctionaid (BLUSA).
Time Frame: Baseline; 2 weeks post BLUSA
Population: Change could only be assessed for 22 participants because 3 participants in the intervention arm dropped out prior to the post assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline | 44.65 (14.42) | 42.78 (13.76)
  2-weeks post BLUSA: number analyzed (Participants) | 22 | 25
  2-weeks post BLUSA | 50.24 (22.52) | 49.41 (15.18)

2. Primary Outcome: Change in Quality of Life
Description: Voice-Related Quality of Life (V-RQOL). It is a 10-item scale with each items 2 - 10 and total score ranges from 20 - 100. Lower scores refers to higher quality of life and Higher scores refer to lower level quality of life.
Time Frame: Baseline; 2 weeks post BLUSA
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline | 26.59 (16.81) | 26.67 (16.72)
  2-weeks post BLUSA: number analyzed (Participants) | 22 | 25
  2-weeks post BLUSA | 42.50 (17.69) | 32.26 (24.90)

3. Secondary Outcome: Speech Intelligibility
Description: The Speech Intelligibility Test has 11 randomly computer generated sentences that patients are asked to read aloud. They are recorded and judged by an unfamiliar listener at a later time. Scores range from 0 - 100 with higher scores indicating greater level of speech intelligibility.
Time Frame: 2 weeks
Population: Only 18 participants in the intervention group were assessed because only 18 of them were able to read the sentences. No data was collected from any participants in the control group for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of intelligible sentences
Arm/Group | Intervention | Control
Number analyzed (Participants) | 18 | 0
percentage of intelligible sentences | 53.1 (25.8) |

4. Secondary Outcome: Level of Independence With Talking Tracheostomy Tube
Description: Participants were asked how independently they thought they could use the tracheostomy tube. Will report the number of participants who indicated some level of independence.
Time Frame: 2 weeks
Population: This outcome was assessed for all 22 participants who completed the intervention arm. No data was collected for any of the participants in control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 22 | 0
Participants | 16 |

5. Secondary Outcome: Patient Satisfaction With a Talking Tracheostomy Tube
Description: Participants were asked how satisfied they were with the tracheostomy tube. Will report the number of participants who indicated some level of satisfaction.
Time Frame: 2 weeks
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 22 | 0
Participants | 9 |

6. Secondary Outcome: Overall Hospital Length of Stay
Description: Measured in days
Time Frame: Time of discharge from the hospital (Approximately 6-8 months)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 25
days | 72.68 (40.94) | 48.84 (27.61)

7. Secondary Outcome: Intensive Care Unit (ICU) Length of Stay
Description: Measured in days
Time Frame: Time of discharge from the ICU (Approximately 6-8 months)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 25
days | 58.12 (36.56) | 39.04 (23.71)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of consent to 2 weeks post intervention.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT02018562/Prot_SAP_000.pdf